CLINICAL TRIAL: NCT07391917
Title: ALExSEM - Hypersensibilité au Liquide séminal : Qualité de Vie ALExSEM - Human Seminal Plasma Allergy: Quality of Life
Brief Title: Human Seminal Plasma Allergy: Quality of Life
Acronym: ALExSEM
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025-A02920-49
Record Dates: First submitted 2026-01-19; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Allergic Reaction
Keywords: seminal fluid; allergy; sexuality; quality of life; Human Seminal Plasma Allergy (HSPA)
MeSH Terms: conditions — Hypersensitivity; Sexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women with HSPA: Measure of quality of life with different questionnaires

SUMMARY:
Human Seminal Plasma Allergy (HSPA) is a rare allergy with localized and/or generalized manifestations following exposure during unprotected sex. Its cause remains undetermined and is certainly underdiagnosed. It is an under-recognized cause of acute or chronic pain related to penetration and vaginal inflammation affecting sexually active women.

To date, no quality-of-life questionnaire specific to this condition exists to demonstrate its impact on the physical, mental, and sexual health of patients.

To try to highlight the suffering of these patients, non-specific sexual quality-of-life questionnaires exist and could be used, such as the "Female Sexual Function Index" (including questions on desire, arousal, and the ability to reach orgasm), but these do not address the sexual impact of psychological distress related to any pathology and do not assess the impact of HSPA-specific symptoms on sexuality. The symptoms of endometriosis can be compared to those of patients with HSPA due to chronic abdominopelvic pain that worsens during sexual intercourse, the psychological impact, and the potential effect on fertility.

A specific questionnaire exists for patients with endometriosis that documents these commonalities: the EHP-30. It is recognized as a specific and sensitive tool for measuring the quality of life of women with endometriosis in routine clinical practice. However, the EHP-30 questionnaire focuses on symptoms that are often chronic and persistent, even outside of sexual intercourse, whereas HSPA is characterized by acute episodes, sometimes spaced out and dependent on exposure to seminal fluid, making the tool less relevant for assessing the quality of life of patients with HSPA.

This study aims to evaluate and compare the measurement of quality of life in patients with HSPA using these different tools and a specific general question in order to describe quality of life in this population. This will also provide evidence to question the value of creating a questionnaire specific to the pathology.

DETAILED DESCRIPTION:
After enrollment and questionnaire collection, relevant medical data are gathered from the medical record (data recorded during the consultation) :

* General data: age, weight/height, number of children, desire for pregnancy, use of assisted reproductive technology, presence of a male dog or cat in the home
* Comorbidities at diagnosis: atopic predisposition, allergies, asthma, eczema, urticaria, chronic rheumatological/urological/gynecological/psychiatric/other conditions
* Characterization of the seminal fluid allergy: date of diagnosis, symptoms, number of partners with whom symptoms have occurred, time to onset of symptoms after exposure, duration of symptoms, results of allergy testing (prick tests, specific IgE, seminal fluid TB test)
* Treatments offered and response (if applicable)
* Outcome: Stability, improvement, worsening, recovery

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Treated at Angers University Hospital for Human Seminal Plasma Allergy during the period of interest (2010-2026)

Exclusion Criteria:

* Objecting to participating in the research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with Human Seminal Plasma Allergy (HSPA)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2026-08-22 (Estimated); Study Completion 2026-08-22 (Estimated)

PRIMARY OUTCOMES:
Overall Quality of life (WHOQOL-BREF) | 1 day
  Measure of overall and domain-specific quality of life using the WHOQOL-BREF questionnaire (26 items).
  Unit of measurement: quality of life scores (overall score and scores for the 4 domains: physical health, psychological health, social relationships, environment), calculated from items rated on a Likert-type scale and converted into continuous scores (items scores between 4 and 20 ; higher scores = better quality of life).
Sexual Quality of life (FSFI) | 1 day
  Measure of sexual quality of life using the Female Sexual Function Index (FSFI) questionnaire.
  Unit of measurement: total FSFI score and scores for individual domains (desire, arousal, lubrication, orgasm, satisfaction, pain), calculated from items rated on a Likert-type scale (higher scores = better sexual function). Total score of 2 to 36.
Quality of life and chronic gynecological condition (EHP30) | 1 day
  Measure of the impact of endometriosis on quality of life using the Endometriosis Health Profile 30 (EHP 30) questionnaire as a reference for the chronic gynecological condition HSPA Unit of measurement: scores for domains (including pain, control and power, emotional well-being, social relationships, and work life), expressed on a scale of 0 to 4. Total score of 0 to 100 (0 = no impact/best quality of life, 100 = maximum impact on quality of life/worst quality of life).
Quality of life and HSPA | 1 day
  Perceived quality of life related to the HSPA is measured using a general question:
  "How would you rate your overall quality of life in relation to your HSPA?" Unit of measurement: score on a numerical scale from 0 to 10 (0 = worst quality of life; 10 = perfect quality of life).

SECONDARY OUTCOMES:
Relationships between the scores | 1 day
  The relationships between the different assessment tools (WHOQOL-BREF, FSFI, sections C to F of the EHP-30, and the general quality of life question) will be explored using Spearman correlations. Correlation coefficients will be visualized as a correlation matrix (corrplot) to identify potential links between the dimensions assessed by the different questionnaires.
Perception of validated questionnaires used | 1 day
  An assessment of the questionnaire's relevance in evaluating the impact of the pathology on quality of life is included at the end of each questionnaire. Responses to these questions are given on a 4-point Likert scale.
  * Is the questionnaire relevant and sufficiently specific to the issues related to HSPA? (0 = Not at all relevant to 3 = Very relevant)
  * Do you feel that certain important dimensions of HSPA are neglected/not addressed? (0 = Strongly disagree to 3 = Strongly agree)
  * Do you think this questionnaire alone is sufficient to highlight the impact of HSPA on your quality of life? (0 = Strongly disagree to 3 = Strongly agree)
  * Do you find some questions and/or sub-scores unnecessary? (0 = Strongly disagree to 3 = Strongly agree)
Population | 1 day
  Describe the characteristics of the population treated at the University Hospital of Angers for HSPA
Risk factors | 1 day
  Explore risk factors associated with the overall quality of life score related to HSPA:
  Current BMI: < 20 kg/m²; 20-29 kg/m²; ≥ 30 kg/m² Age: 18-35 years; 35-50 years; > 50 years Number of biological children Desire for pregnancy History of eczema History of respiratory allergies and/or asthma

CONTACTS AND LOCATIONS:
Overall Officials: Martine MORISSET, Dr, Principal Investigator — University Hospital of Angers
Locations (1):
- Sandra MERZEAU, Angers, France